CLINICAL TRIAL: NCT03980158
Title: Change in Tongue Strength and Fatigue After Implantation of Upper Airway Stimulation System
Brief Title: Change in Tongue Strength and Fatigue After Upper Airway Stimulation Therapy
Status: Completed | Type: Observational
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: 425/17S
Record Dates: First submitted 2019-05-26; First posted 2019-06-10 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Obstructive Sleep Apnea of Adult

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Upper airway stimulation group
- OSA group with conservative / no treatment
- Test group without OSA

SUMMARY:
Upper airway stimulation (UAS) is an effective surgical alternative for patients with obstructive sleep apnea (OSA) who fail continuous positive airway pressure (CPAP) therapy. This stimulation could lead to alterations in tongue strength and fatigability which could alter treatment outcome. The aim of the study is to investigate if UAS alters tongue strength and fatigability.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* upper airway stimulation group: Upper airway stimulation system implanted at least 4 weeks ago
* OSA group: OSA confirmed by 18-channel inpatient overnight polysomnography (PSG)
* test group: No medical history for OSA and Epworth Sleepiness Scale (ESS) below 11

Exclusion Criteria:

* history of a neuromuscular disorder
* previous tongue surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of three groups: the first group comprises of patients that have been implanted with selective hypoglossal nerve stimulation system (Inspire II Upper Airway Stimulation System, Inspire Medical Systems, Maple Grove, USA). The second group consists of confirmed OSA patients either being treated conservatively or without treatment. The test group consists of participants with no medical history for OSA and Epworth Sleepiness Scale (ESS) below 11.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-11-16 (Actual); Study Completion 2018-11-16 (Actual)

PRIMARY OUTCOMES:
Tongue protrusion strength | Up to 60 months after implanation
  Tongue protrusion strength (peak pressure in kPa)
Tongue fatigability | Up to 60 months after implanation
  Time to task failure during 50% of peak pressure contraction in seconds

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ear Nose Throat, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wirth M, Unterhuber D, von Meyer F, Hofauer B, Ott A, Edenharter G, Eckert DJ, Heiser C. Hypoglossal nerve stimulation therapy does not alter tongue protrusion strength and fatigability in obstructive sleep apnea. J Clin Sleep Med. 2020 Feb 15;16(2):285-292. doi: 10.5664/jcsm.8184. Epub 2020 Jan 13. PMID 31992396